CLINICAL TRIAL: NCT07359209
Title: Study on the Mechanism s of Berberine Improving Cognitive Impairments in Schizophrenia Based on "Gut m Icrobiota-gut-brain"Axis
Brief Title: Berberine Improving Cognitive Impairments in Schizophrenia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Anding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBR-SCH-2023
Record Dates: First submitted 2023-07-22; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia Therapeutics
Keywords: schizophrenia; berberine; cognitive symptoms; Intestinal flora
MeSH Terms: conditions — Schizophrenia; Neurobehavioral Manifestations | interventions — Berberine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine group (Experimental)
  Interventions: Drug: Berberine
- control group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Berberine — Berberine 300mg#three times a day# plus any stable antipsychotic drug
  Other Names: stable antipsychotic
  Arms: berberine group
Drug: Placebo — The placebo were matched to Berberine in shape, smell and colour and tablets were sealed in identical bottles
  Other Names: stable antipsychotic
  Arms: control group

SUMMARY:
The study was a 12-week, randomized, double-blind, placebo-controlled trial. Berberine (300 mg, three times a day) has been used as an auxiliary treatment on the basis of stable antipsychotic treatment. All participants were randomly divided into two groups.Any stable antipsychotic + berberine(BBR) or any stable antipsychotic +placebo. Positive and Negative Syndrome Scale (PANSS) has been used for psychiatric symptoms. MATRICS Consensus Cognitive Battery（MCCB）has been used for cognitive symptoms. The treatment Emergent Symptom Scale(TESS) has been used for evaluate adverse effects. Plasma Metabolomics, Inflammatory Factors, BDNF, fecal Macrogene Sequencing, and fecal Metabolomics were obtained at 0, 4,8 ,12weeks.

DETAILED DESCRIPTION:
Plasma Metabolomics, Inflammatory Factors, BDNF, fecal Macrogene Sequencing, and fecal Metabolomics were obtained at 0, 4,8 ,12weeks.

Inflammatory factors:C-reaction protein(CRP),Interleukine-1 beta(IL-1β), Interleukine-6 (IL-6), Tumor necrosis factor-α (TNF-α).

ELIGIBILITY:
Inclusion Criteria:

* Individuals who aged 18 to 60 years
* Meet the diagnosis of schizophrenia according to DSM-V
* Treatment with stable Antipsychotic ≥ 3 months, and the drug dose was not adjusted 1 month before enrollment
* The total score of the Positive and Negative Syndrome Scale (PANSS) ≤ 70 points, with scores of item delusion, conceptual confusion, hallucination, and excitement ≤ 4 points
* The MATRICS Conscience Cognitive Battery for Schizophrenia,MCCB) scoring defect score ≥ 3 points
* Gender unlimited
* Sign the informed consent form

Exclusion Criteria:

* Individuals who with diagnosis of other psychiatric disorders except schizophrenia according to DSM-V
* Refused to provide informed consent
* Significant medical illnesses including uncontrolled hypertension, diabetes, seizure disorder, severe cardiovascular, cerebrovascular, pulmonary, or thyroid diseases
* Currently on anti-inflammatory or immunosuppressant medication including oral steroids and history of chronic infection (including tuberculosis, HIV and hepatitis), malignancy, organ transplantation, blood dyscrasia, central nervous system demyelinating disorder, and any other known autoimmune or inflammatory condition.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2028-07-23 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Changes of cogination symptoms | changes within 0,4,8,12weeks
  MCCB is a standardized measurement tool for assessing cognitive function in schizophrenia. There are 9 subtests, which mainly assess 7 cognitive domains, including information processing speed, attention/alertness, Working memory, word learning, visual memory, reasoning and problem solving, and social cognition. After the evaluation is completed, the MCCB rough score is converted into the total score T score obtained after correction for age, gender, years of education, and untreated period. The T score is then converted into a defect score, with T scores ≥ 40, 35-39, 30-34, 25-29, 20-24, and ≤ 19 corresponding to defect scores 0, 1, 2, 3, 4, and 5, respectively. Among them, 1 represents mild defects, 2 represents mild to moderate defects, 3 represents moderate defects, 4 represents moderate to severe defects, and 5 represents severe defects. In this study, a defect score of ≥ 3 was used as the boundary for significant cognitive impairment.

SECONDARY OUTCOMES:
Changes of CRP | changes within 0, 4, 8, 12weeks
  The concentration of C-reactive protein (CRP) is measured in venous blood. CRP is an acute-phase reactant protein synthesized by the liver, primarily functioning to recognize and clear pathogens or damaged cells. It plays a crucial role in inflammatory responses, infection surveillance, and disease monitoring.
Changes of Plasma Metabolomics(PM) | changes within 0, 12weeks
  Collected and stored plasma samples were registered in the MetLIMS software, including relevant sample information. Subsequently, these samples underwent mass spectrometry-based detection and quantification. Each sample was divided into two aliquots for analysis: the first aliquot was subjected to Flow Injection Analysis (FIA) mode for signal acquisition, and the second aliquot was analyzed using Liquid Chromatography-Mass Spectrometry (LC-MS) mode. The resultant data were imported into the Biocrates MetIDQ™ software for the precise calculation of analyte concentrations and comprehensive data evaluation. Further analysis was conducted utilizing the MetaboAnalyst 5.0 platform, along with resources such as the KEGG database, to identify significant metabolites and explore associated metabolic pathways.
Changes of IL-1β | changes within 0,4,8,12weeks
  The levels of IL-1β has been obtained at 4 point intervals: 0, 4, 8,12 weeks
Changes of IL-6 | changes within 0,4,8,12weeks
  The levels of IL-6 has been obtained at 4 point intervals: 0, 4, 8 ,12weeks
Changes of TNF-α | changes within 0,4,8,12weeks
  The levels of TNF-α has been obtained at 4 point intervals: 0, 4, 8 ,12weeks
Changes of BDNF | changes within 0,4,8,12weeks
  The levels of BDNF has been obtained at 4 point intervals: 0, 4, 8,12 weeks
Changes of Fecal Macrogene Sequencing(FMS) | changes within 0, 12weeks
  Total genomic DNA was extracted from patient fecal samples and subjected to quality control. Qualified DNA was then randomly fragmented to approximately 350 bp using a Covaris ultrasonic disruptor to generate libraries, which were quantified by Qubit and qPCR. Following library QC, pooled libraries were sequenced on an Illumina NovaSeq platform (PE150). Raw sequencing data underwent quality control, followed by assembly and gene prediction to construct a non-redundant gene set. Genes were then annotated for taxonomic and functional classification and abundance statistics were computed. Statistical analyses, including similarity clustering, group ordination, and differential comparisons, were performed on samples and sample groups.
Changes of Fecal Metabolomics(FM) | changes within 0, 12weeks
  Collected and stored patient fecal samples were registered in the MetLIMS software, including relevant sample information. Subsequently, these samples underwent mass spectrometry-based detection and quantification. Each sample was divided into two aliquots for analysis: the first aliquot was subjected to Flow Injection Analysis (FIA) mode for signal acquisition, and the second aliquot was analyzed using Liquid Chromatography-Mass Spectrometry (LC-MS) mode. Data Processing and Pathway Analysis: The resultant data were imported into the Biocrates MetIDQ™ software for the precise calculation of analyte concentrations and comprehensive data evaluation. Further analysis was conducted utilizing the MetaboAnalyst 5.0 platform, along with resources such as the KEGG database, to identify significant metabolites and explore associated metabolic pathways.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Anding Hospital, Tianjin, China